CLINICAL TRIAL: NCT03376698
Title: A Randomized, Double-blind, Placebo-controlled Phase II Trial to Evaluate the Dose-dependent Effect of Colchicine on Inflammatory Response and Endothelial Function in Type 2 Diabetic Patients With Coronary Artery Disease and Leukocyte Activation
Brief Title: Dose-finding Study of Colchicine in Type 2 Diabetic Patients With Coronary Artery Disease
Acronym: DRC-04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of the Ryukyus (Other)
Responsible Party: Principal Investigator, Shinichiro Ueda, Professor, University of the Ryukyus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1195
Record Dates: First submitted 2017-10-23; First posted 2017-12-18 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Colchicine; Diabetes Mellitus, Type 2; Coronary Artery Disease; White Blood Cell; Inflammation; Diarrhea
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Inflammation; Diarrhea | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Colchicine 0.5 mg (Active Comparator)
  Interventions: Drug: Colchicine 0.5 mg
- Colchicine 0.25 mg (Active Comparator)
  Interventions: Drug: Colchicine 0.25 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 mg — oral administration of Colchicine 0.5 mg once daily for 12 weeks
  Arms: Colchicine 0.5 mg
Drug: Colchicine 0.25 mg — oral administration of Colchicine 0.25 mg once daily for 12 weeks
  Arms: Colchicine 0.25 mg
Drug: Placebo — oral administration of Placebo once daily for 12 weeks
  Arms: Placebo

SUMMARY:
This study is designed to investigate dose-dependent effects of low dose colchicine on inflammatory responses, endothelial function in type 2 diabetic patients with coronary artery disease and leukocyte activation. This study also tested the relationship between doses and safety issue such as incidence of diarrhea. Eligible patients will be randomly allocated to three treatment group: colchicine at 0.5mg per day, 0.25mg per day or placebo for 12 weeks in a double blind , parallel group design. High sensitive-CRP at 4 weeks as primary end point and flow mediated vasodilatation at 12 weeks as the secondary end point will be measured.

DETAILED DESCRIPTION:
Mortality rate in Japanese coronary artery disease (CAD) patients has been deemed the lowest among developed countries for the long time. However, cohort study of the investigators based on the registry of 8000 patients with CAD and type 2 diabetes has shown that cardiovascular mortality of such patients even under the optimized standard therapy and relatively intensive control of risk factors was higher than the investigators thought. Given substantial experimental evidence suggesting roles of inflammation as a key player in the development of atherosclerosis and significant association of enhanced inflammatory reaction and cardiovascular events in registry-based cohort of the investigators, the investigators are planning of phase 3 trial of colchicine, which is an ancient anti-inflammatory drug, for the regulatory approval as a drug preventing of cardiovascular events in diabetic CAD patients with enhanced inflammatory reaction. To develop appropriate study protocol of phase 3 trial, a dose-finding study is apparently warranted since our pharmacokinetics study and pharmacokinetics /pharmacodynamics study showed that colchicine stays in leukocytes with a long half life being more than 40 hours and showed consistent inhibition of leukocyte activation for more than 48 hours. In terms of safety issue, 0.5mg of colchicine, which has been frequently used in several cardiovascular trials, is associated with high incidence of diarrhea. As dose-dependency is assumed regarding diarrhea, a dose finding study for safety issue is also needed. The investigators, thus, conduct a double-blind randomized controlled trial to investigate dose-dependent effects on inflammatory responses using highly sensitive-CRP as an indicator, endothelial function using FMD, and incidence of diarrhea comparing once daily oral administration of 0.5 mg, 0.25 mg of colchicine and placebo for 12 weeks in CAD patients with type 2 diabetes mellitus and leukocyte activation. The investigators focus on patients with type 2 diabetes and leukocyte activation among CAD patients for regulatory approval because it is likely that such patients are at highest risk and respond well to colchicine.

ELIGIBILITY:
Inclusion Criteria:

* The subjects in this trial must have all of the following criteria.

  1. Patients with type 2 diabetes mellitus with coronary artery disease(*1) with increased inflammatory response(*2).

     * 1:"Type 2 diabetes" mellitus is diagnosed by criteria according to The Japan Diabetes Society. "Coronary artery disease" is defined as having equal to or greater than 75% stenosis in coronary angiography, history of acute coronary syndrome, and history of coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI).
     * 2:"Increased inflammatory response" is defined as follow; White blood cell levels at confirmation tests of eligibility is equal to or greater than 7000 /μL.
  2. Patients aged 20 years and older
  3. In female subjects who had possibility of pregnancy and male subjects who had female partner who had possibility of pregnancy and not undergone a contraceptive surgery(*3), patients with consent of performing optimal contraception from starting study drug to 90 days from final taking.

     * 3: Male subjects who had undergone a contraceptive surgery are defined as elapsing for at least one year after vasectomy and having a certification of no sperm at ejaculation.
  4. After receiving sufficient explanation for the participation of this study, patients who wrote document of informed consent by the patient's free will with sufficient understanding.

Exclusion Criteria:

* The subjects who conflict with at least one of the following criteria are exclude from this trial.

  1. Patients with prior hypersensitivity to Colchicine.
  2. Patients with taking Colhicine presently or to 30 days before confirmation tests of eligibility.
  3. Patients with liver cirrhosis
  4. Patients with clinical cholestasis.
  5. Patients with decreasing renal function (eGFR < 30 mL/min/1.73m2) at confirmation tests of eligibility.
  6. Patients with active malignancy.
  7. Patients taking drugs that are indicated as "combined caution" in the package insert of Colchicine as a drug which may interact with Colchicine. 1. Drugs inhibiting cytochrome P450 drug-metabolizing enzyme

     1. Strong Inhibitor Atazanavir, Clarithromycin, Indinavir, Itraconazole, Nelfinavir, Ritonavir, Saquinavir, Darunavir, Telithromycin, Telaprevir, Preparation including Cobicistat
     2. Moderate Inhibitor Amprenavir, Aprepitant, Diltiazem, Erythromycin, Fluconazole, Fosamprenavir, Verapamil 2. P-glycoprotein inhibitor Ciclosporin
  8. Patients taking Amiodarone or Quinidine.
  9. Patients with infectious or inflammatory disease at confirmation tests of eligibility.
  10. Current smoker
  11. Patients with pregnancy, possible pregnancy, on breast-feeding or who wish to become pregnant during trial. (The female subjects who had possibility of pregnancy receive a pregnancy test.)
  12. Patients registered in other clinical trials presently or within 30 days before acquisition consent of this trial.
  13. Patients whom physician in charge considered inappropriate for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in serum high-sensitivity CRP (mg/dl) | 4 weeks

SECONDARY OUTCOMES:
Change in serum high-sensitivity CRP (mg/dl) | 12 weeks
Change in Flow Mediated Dilatation (%) | 12 weeks
Change in adhesive ability of white blood cell (number/field of view) | 4 weeks
Change in time through the microchannel of white blood cell (sec) | 4 weeks
Change in plasma myeloperoxidase level (ng/ml) | 4 and 12 weeks

OTHER OUTCOMES:
Cardiovascular events | 12 weeks
  death, myocardial infarction, stroke, hospitalization due to worsening heart failure, unstable angina
Adverse events | 12 weeks
Side effect | 12 weeks
Diarrhea | 12 weeks
  especially notable adverse event
Concentration of colhicine in plasma (ng/ml) | 12 weeks
  feasible facility only
Concentration of colhicine in white blood cell (ng/1*10^9 cells) | 12 weeks
  feasible facility only

CONTACTS AND LOCATIONS:
Overall Officials: Shinichiro Ueda, PhD, Principal Investigator — blessyou@med.u-ryukyu.ac.jp
Locations (5):
- Japan (5):
  - Hiroshima University Hospital, Hiroshima
  - Kitasato University Hospital, Kanagawa
  - Urasoe Sogo Hospital, Okinawa
  - Dokkyo Medical University Nikko Medical Center, Tochigi
  - Showa University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided